CLINICAL TRIAL: NCT03346031
Title: Assessment of the Effect of Music Therapy on Analgesia and Oxidative Stress Parameters in Anesthetized Oocyt Pickup Patients
Brief Title: The Effect of Music Therapy on Analgesia and Oxidative Stress Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Yavuz Orak, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017/12-14
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-07

CONDITIONS: Infertility; Anesthesia
Keywords: music therapy, pain, oxidative stress parameters
MeSH Terms: conditions — Infertility; Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (No Intervention): Group 1 is control group that does not listen to music
- Music Therapy Group 2 (Active Comparator): Group 2 is the group listening to preoperative music
  Interventions: Procedure: music therapy
- Music Therapy Group 3 (Active Comparator): Group 3 is the preoperative and peroperative music listening group (continuous)
  Interventions: Procedure: music therapy

INTERVENTIONS:
Procedure: music therapy — patients will listen to music with an MP3 headset
  Arms: Music Therapy Group 2; Music Therapy Group 3

SUMMARY:
Music has been used in the treatment of patient since the time Plato, Hippocrates and Alpharabius were alive. It is used by music therapists to help patients' social, physical, emotional, psychological and spiritual needs. In a study conducted, it was seen that music has a positive effect on pain, anxiety, depression, shortness of breath, mood, face expression and speech. Our aim is to evaluate the analgesic consumption of music therapy during egg collection applications and to compare the parameters of oxidative stress in blood and follicular fluid.

DETAILED DESCRIPTION:
Patients were randomly allocated into 3 groups. Group 1 is control group. Group 2 is Classical Turkish Music group. Group 3 will be organized as a group listening continuously (Preoperative and peroperative) Classical Turkish Music (Acemaşiran Makam). Voluntary patients, patients without hearing problems, patients between the ages of 18 and 40, and patients without music phobia will be included in the study. Patients who do not want to participate in the study, patients with hearing problems, and patients outside the 18-40 age range will not be included in the study. Once the Control group has been taken to the patient's room, the vessel way will be prepared for operation and will be kept waiting for one hour. Then blood will be taken to evaluate the oxidative stress parameters (Superoxide Dysmotase, Catalase, Glutathione Peroxidase, Myeloperoxidase, Malondialdehyde, Nitric Oxide, Thiol Disulfide levels) and taken to the operation room. Group 2 patients will be taken to the patient's rest room and will listen to music with an MP3 headset for 1 hour. Patient's blood will be taken to assess the oxidative stress parameters and taken to the operation room. Group 3 will listen Turkish Classical Music for 1 hour in patient room, vein path will be opened, Patient's blood will be taken with the aim of evaluating oxidative stress parameters and taken to the operation room. The patients will listen to music throughout the operation. All patients included in the study (Gr.1, Gr.2, Gr.3 patients) will use remifentanil 0.5 mcg / kg, propofol 1 mg / kg on induction after taken to the operating table. Hemodynamics (Systolic Blood Pressure, Diastolic Blood Pressure, Heart Rate, Oxygen Saturation, Mean arterial pressure) and body movements of all patients included in the study will be recorded. Additional anesthesia and analgesia needs will be recorded during the operation at 1,3,5,7,10,15 minutes. Blood and follicle fluid will be taken with the aim of comparing the values of Oxidative Stress Parameters in blood and follicular fluid at the end of the operation of all the patients in the three groups included in the study. Hemodynamics follow-up and pain follow-ups will be recorded at 1,5,15,30, and 60 minutes in the postoperative resting rooms of the patients after the operation. VAS will be used for pain recording. The analgesic needs of the patients will be met. Non-steroidal anti-inflammatory drugs will be administered to patients for postoperative analgesia. The pre-and post-operative oxidative stress parameters in patients blood will be compared and the oxidative stress parameter values of the follicular fluid of the patients after the operation will be compared in the three groups.

ELIGIBILITY:
Inclusion Criteria:

1.Voluntary patients

1. patients without hearing problems
2. patients between the ages of 18 and 40
3. patients without music phobia

Exclusion Criteria:

1. Patients with hearing problems.
2. Patients older than 18 years and older than 40 years
3. Patients who do not want to participate in the trial
4. Patients with music phobia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers with the music therapy | Change from baseline at 1 hour
  To evaluate the impact on the circulating levels of Catalase ü/ml,Glutathione Peroxidase ü/ml, Myeloperoxidase ü/ml, Malondialdehyde nmol/ ml, Nitric Oxide umol/ L, Thiol Disulfide

SECONDARY OUTCOMES:
Pain Scores | 1 minute,5 minute,15 minute,30 minute, 60 minute of pain level after operation
  VAS (Visual analog scale) Score. from 1 to 10 , 0: No pain, 10: 10 pain that can not be tolerated
Hemodynamics and oxygen follow-up | During the operation, 1 minute, 3 minutes, 5 minutes, 7 minutes, 10 minutes, 15 minutes.Each unit will be evaluated separately within itself
  Systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate,
Hemodynamics and oxygen follow-up | after the operation in 1 minute, 5 minutes, 15 minutes, 30 minutes, 60 minutes.Each unit will be evaluated separately within itself
  Systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate,

CONTACTS AND LOCATIONS:
Overall Officials: yavuz orak, md, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University Faculty of Medicine, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No